CLINICAL TRIAL: NCT06684223
Title: Analysis of Surgical and Oncologic Outcomes After Compete Mesocolic Excision or Non-complete Mesocolic Excision for Right-Sided Colon Cancer
Brief Title: Analysis of Surgical and Oncologic Outcomes After Complete Mesocolic Excision or Non-complete Mesocolic Excision for Right-Sided Colon Cancer
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Korea University Anam Hospital (Other); Kyungpook National University Chilgok Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, In Ja Park, Professor, Asan Medical Center
Other Study IDs: mD3 domestic
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Colon Cancer; Laparoscopic Colon Surgery; Lymph Node Dissection; Robotic Surgical Procedures
Keywords: colon cancer; right hemicolectomy; laparoscopic colectomy; complete mesocolic excision; lymph node dissection; robotic colectomy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who underwent laparoscopic or robotic right hemicolectomy with modifiedD3 from 2013 to 2020: Patients who underwent laparoscopic or robotic right hemicolectomy with modified D3 lymphadenectomy from 2013 to 2020 in 4 centers
- Patients who underwent laparoscopic or robotic right hemicolectomy with CME from 2013 to 2020: Patients who underwent laparoscopic or robotic right hemicolectomy with Complete mesocolic excision from 2013 to 2020 in 4 centers

SUMMARY:
The goal of this observational study is to investigate the efficacy and safety of a modified D3 lymphadenectomy approach compared to Complete Mesocolic Excision (CME) in patients with right-sided colon cancer. The main question it aims to answer is:

Does a modified D3 approach improve disease-free survival (DFS) in patients with Stage I-III right-sided colon cancer who undergo right-sided colectomy, without increasing surgical complications compared to CME?

Patients with right-sided colon cancer, Stage I-III, who undergo either modified D3 lymphadenectomy or CME as part of their standard treatment, will have their DFS, complications, bleeding volume, number of lymph nodes harvested, and stage distribution compared over a follow-up period. This study ultimately aims to determine the optimal surgical approach for maximizing oncologic outcomes in right-sided colon cancer.

DETAILED DESCRIPTION:
This observational, population-based, cohort study was conducted following the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines. Approval was obtained from the institutional review board (IRB) of the primary institution and the ethics committees of each participating institution in the Republic of Korea. Given that the study utilized anonymized data retrospectively, the need for informed consent was waived.

The study aimed to evaluate the efficacy and safety of modified D3 lymphadenectomy compared to Complete Mesocolic Excision (CME) in patients with right-sided colon cancer. Patients with right-sided colon cancer who underwent laparoscopic or robotic right hemicolectomy from 2013 to 2020 were included. Patients were classified into those who received modified D3 lymphadenectomy or CME, and the study assessed disease-free survival (DFS), surgical complications, bleeding volume, lymph node yield, and stage distribution.

Data collection was carried out at multiple tertiary medical centers across the Republic of Korea, ensuring a broad representation of patient demographics and clinical practices. The participating institutions included Asan Medical Center, Korea University Anam Hospital, Severance Hospital, and Kyungpook National University Chilgok Hospital. These centers vary in location and size, enhancing the study's generalizability within the context of right-sided colon cancer management in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic or robotic right hemicolectomy from 2013 to 2020
* Patients who received curative right hemicolectomy with lymphadenectomy

Exclusion Criteria:

* Familial adenomatous polyposis (FAP)
* Hereditary non-polyposis colon cancer (HNPCC)
* Patients with inflammatory bowel disease
* Patients with synchronous malignancies in other organs
* Patients with non-adenocarcinoma histology of colon cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients who underwent laparoscopic or robotic right hemicolectomy from 2013 to 2020 at four institutions: Asan Medical Center, Kyungpook National University Chilgok Hospital, Korea University Anam Hospital, and Yonsei University Severance Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3787 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | Outcome measures will be assessed at 5 years post-surgery.
  Recurrence-Free Survival (RFS) between patients who underwent modified D3 and CME procedures from 2013 to 2020.

SECONDARY OUTCOMES:
Comparison of complication rates between modified D3 and complete mesocolic excision | The outcomes will be assessed to determine if any events occurred post-surgery up to October 2024
  This study will compare the complication rates between modified D3 (mD3) lymphadenectomy and Complete Mesocolic Excision (CME).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No